CLINICAL TRIAL: NCT00777153
Title: A Phase III, Randomised, Parallel Group, Multi-Centre Study in Recurrent Glioblastoma Patients to Compare the Efficacy of Cediranib [RECENTIN™, AZD2171] Monotherapy and the Combination of Cediranib With Lomustine to the Efficacy of Lomustine Alone
Brief Title: Cediranib in Combination With Lomustine Chemotherapy in Recurrent Glioblastoma
Acronym: REGAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D8480C00055
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Glioblastoma
Keywords: Cancer; Tumour; Advanced Solid Tumour; GBM; Glioblastoma
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — cediranib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cediranib 30mg (Experimental): Cediranib 30mg
  Interventions: Drug: Cediranib
- Cediranib 20mg + lomustine (Other): Cediranib 20mg + lomustine
  Interventions: Drug: Cediranib; Drug: Lomustine Chemotherapy
- Lomustine and Placebo Cediranib (Active Comparator): Lomustine and Placebo Cediranib
  Interventions: Drug: Lomustine Chemotherapy; Drug: Placebo Cediranib

INTERVENTIONS:
Drug: Cediranib — 30 mg/day, oral, until progression
  Arms: Cediranib 30mg
Drug: Cediranib — 20 mg/day, oral, until progression
  Arms: Cediranib 20mg + lomustine
Drug: Lomustine Chemotherapy — 110 mg/m2 / Q6W, oral, until progression
  Arms: Cediranib 20mg + lomustine; Lomustine and Placebo Cediranib
Drug: Placebo Cediranib — Oral, until progression
  Arms: Lomustine and Placebo Cediranib

SUMMARY:
The purpose of this study is to see how effective cediranib is in treating a brain tumour called recurrent glioblastoma. Two drugs are being tested in this study. Lomustine is an approved oral chemotherapy that belongs to the class of drugs called alkylating agents. Cediranib is a new drug that has not yet been approved for this disease. This study will compare the use of lomustine with cediranib, cediranib alone or lomustine with placebo ("inactive substance") to see whether the combination or cediranib alone will be more effective than the chemotherapy alone (lomustine) in preventing the growth of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of recurrent glioblastoma
* Life expectancy ≥ 12 weeks
* Received only one prior systemic chemotherapy regimen and this regimen must contain temozolomide

Exclusion Criteria:

* Patients on enzyme-inducing anti-epileptic drugs within 3 weeks prior to randomisation
* Poorly controlled hypertension
* Previous anti-angiogenesis (eg bevacizumab, sorafenib, sunitinib) therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Tracy Batchelor, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (62):
- United States (21):
  - Research Site, Birmingham, Alabama
  - Research Site, Pheonix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Amherst, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
- Australia (6):
  - Research Site, Camperdown
  - Research Site, Heidelberg
  - Research Site, Nedlands
  - Research Site, Parkville
  - Research Site, St Leonards
  - Research Site, Woodville
- Research Site, Graz, Austria
- Belgium (4):
  - Research Site, Brussels (Anderlecht)
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Leuven
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Liberec, Czechia
- France (6):
  - Research Site, Bobigny
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Germany (11):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Nordhausen
  - Research Site, Regensburg
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Rotterdam
  - Research Site, The Hague
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

REFERENCES:
- [Derived] Batchelor TT, Mulholland P, Neyns B, Nabors LB, Campone M, Wick A, Mason W, Mikkelsen T, Phuphanich S, Ashby LS, Degroot J, Gattamaneni R, Cher L, Rosenthal M, Payer F, Jurgensmeier JM, Jain RK, Sorensen AG, Xu J, Liu Q, van den Bent M. Phase III randomized trial comparing the efficacy of cediranib as monotherapy, and in combination with lomustine, versus lomustine alone in patients with recurrent glioblastoma. J Clin Oncol. 2013 Sep 10;31(26):3212-8. doi: 10.1200/JCO.2012.47.2464. Epub 2013 Aug 12. PMID 23940216
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=425&filename=CSR-D8480C00055.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 423 patients were enrolled in to the study but did not start the study. They did not go on to be randomized.
Pre-assignment Details: Randomised=Full Analysis Set (ITT): Cediranib 30 mg=131, Cediranib 20 mg + Lomustine=129, Placebo + Lomustine=65; ITT with measurable disease at baseline (based on site review): Cediranib 30 mg=115, Cediranib 20 mg + Lomustine=112, Placebo + Lomustine=55; Safety Set: Cediranib 30 mg=128, Cediranib 20 mg + Lomustine=123, Placebo + Lomustine=64
Groups:
- Cediranib 30mg: Cediranib 30mg/Day
- Cediranib 20mg + Lomustine 110mg: Cediranib 20mg/Day + Lomustine 110mg/m2/Day
- Lomustine 110mg: Lomustine 110mg/m2/Day + Placebo cediranib
Period: Overall Study
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg
Started | 131 | 129 | 65
Completed | 41 | 46 | 28
Not Completed | 90 | 83 | 37
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 85 | 73 | 33
Not completed — Withdrawal by Subject | 3 | 4 | 3
Not completed — Incorrect enrol/elig crit not fulfilled | 1 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg | Total
Number analyzed (Participants) | 131 | 129 | 65 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Informed Consent
  years | 53.4 (11.81) | 53.7 (10.78) | 52.0 (13.09) | 53.3 (11.67)
Gender [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 46 | 44 | 24 | 114
    Male | 85 | 85 | 41 | 211

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: For patients with measurable disease at entry (at least one lesion that has a shortest diameter
  ≥10 mm at baseline on 2 axial slices), PFS will be defined as the earliest time that:
  1. The sum of the products of the largest perpendicular diameters of contrast enhancement for all lesions has increased by a greater than or equal to 25% in comparison to the nadir scan as long as the shortest diameter is ≥15 mm. If the dose of steroids has been reduced within the 10 days prior to the scan being conducted, progression will be based on a follow-up scan performed after the dose of steroids has been stabilized for 10 days.
  2. The patient has died from any cause.
  3. A new lesion is detected that is outside the original tumor volume and has a shortest diameter ≥10 mm.
Time Frame: Baseline at 6 weeks and then every 6 weeks to discontinuation
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Cediranib 20mg+ Lomustine 110mg: Cediranib 20mg/Day + Lomustine 110mg/m2/Day
Arm/Group | Cediranib 30mg | Cediranib 20mg+ Lomustine 110mg | Lomustine 110mg
Number analyzed (Participants) | 131 | 129 | 65
Days | 92 [80 to 128] | 125 [83 to 201] | 82 [42 to 168]

2. Secondary Outcome: Overall Survival (OS)
Description: Number of months from randomisation to the date of death from any cause
Time Frame: Baseline through to date of death up to 25th April 2010
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg
Number analyzed (Participants) | 131 | 129 | 65
Months | 8.0 [4.1 to 14.5] | 9.4 [6.2 to 14.5] | 9.8 [4.9 to NA] — Third quartile has not been reached.

3. Secondary Outcome: Response Rate
Description: An individual visit response of PR was defined as a greater than or equal to 50% reduction in the sum of the products of the largest perpendicular diameters of contrast enhancement for all lesions compared to baseline as long as the steroid dose has not been increased within the previous 10 days and no new lesions are present.
  An individual visit response of CR was defined as the complete disappearance of all tumor on MRI scan.
Time Frame: Baseline at 6 weeks and then every 6 weeks to discontinuation
Population: Patients are only included in the analysis if they have measurable disease at baseline based on central.
Measure: Number; unit: Participants
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg
Number analyzed (Participants) | 118 | 122 | 56
Participants | 18 | 21 | 5

4. Secondary Outcome: Alive and Progression Free Rate at 6 Months (APF6)
Description: Proportion of patients alive and progression free at 6 months (based on central review) as estimated from Kaplan-Meier techniques. Values are percentages.
Time Frame: 6 Months
Measure: Number; unit: % of patients alive and progression free
Groups:
- Cediranib 20mg + Lomustine 100mg: Cediranib 20mg/Day + Lomustine 110mg/m2/Day
- Lomustine 100mg: Lomustine 110mg/m2/Day + Placebo cediranib
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 100mg | Lomustine 100mg
Number analyzed (Participants) | 131 | 129 | 65
% of patients alive and progression free | 16.2 | 34.5 | 24.5

5. Secondary Outcome: Daily Steroid Dose
Description: The mean steroid dosage prior to treatment will be considered as the patient's baseline. The percent change in average daily steroid dosage from baseline is calculated by following formula: PC = (md - bm)/bm*100; where PC is the percent change in average daily steroid dosage from baseline; md the mean daily steroid dosage recorded from the first day of therapy to progression; and bm the baseline mean.
Time Frame: Baseline to the date of first documented progression or date of death or study discontinuation, whichever came first, assed up to 2014-April-25
Measure: Number; unit: percentage of change
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg
Number analyzed (Participants) | 61 | 68 | 26
percentage of change | -17.6 | -1.8 | 36.6

6. Secondary Outcome: Steroid Free Days
Description: Number of days known not to have used any steroids prior to progression
Time Frame: Baseline to the date of first documented progression or date of death or study discontinuation, whichever came first, assessed up to 2014-April-25
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Cediranib 20mg + Lomustine 119mg: Cediranib 20mg/Day + Lomustine 110mg/m2/Day
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 119mg | Lomustine 110mg
Number analyzed (Participants) | 128 | 123 | 64
Days | 75.8 (110.1) | 74.8 (91.7) | 92.3 (122.0)

ADVERSE EVENTS:
Description: Adverse events are assessed on all patients who meet the Safety set criteria i.e. all patients who were randomized and received at least one dose of study drug.
  Safety Set: Cediranib 30 mg=128, Cediranib 20 mg + Lomustine=123, Placebo + Lomustine=64
Arm/Group | Cediranib 30mg | Cediranib 20mg + Lomustine 110mg | Lomustine 110mg
Serious Adverse Events (participants affected / at risk) | 55/128 | 45/123 | 26/64
Other Adverse Events (participants affected / at risk) | 124/128 | 120/123 | 61/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30mg (N=128) | Cediranib 20mg + Lomustine 110mg (N=123) | Lomustine 110mg (N=64)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 8 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Addison's Disease (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 2 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Feeding Tube Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 11 | 3 | 2
Grand Mal Convulsion (Nervous system disorders) | 3 | 1 | 0
Hemiparesis (Nervous system disorders) | 3 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 2 | 0
Ischaemic Stroke (Nervous system disorders) | 2 | 0 | 0
Neurological Symptom (Nervous system disorders) | 0 | 0 | 2
Partial Seizures (Nervous system disorders) | 1 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebral Cyst (Nervous system disorders) | 0 | 0 | 1
Cerebral Haematoma (Nervous system disorders) | 0 | 0 | 1
Cerebral Venous Thrombosis (Nervous system disorders) | 0 | 1 | 0
Complex Partial Seizures (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Intracranial Pressure Increased (Nervous system disorders) | 0 | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Neurological Decompensation (Nervous system disorders) | 1 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0
Sinus Headache (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Speech Disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 2 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Personality Change (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 4 | 1
Hypertension (Vascular disorders) | 3 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 30mg (N=128) | Cediranib 20mg + Lomustine 110mg (N=123) | Lomustine 110mg (N=64)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 69 | 28
Neutropenia (Blood and lymphatic system disorders) | 2 | 28 | 8
Leukopenia (Blood and lymphatic system disorders) | 2 | 25 | 11
Anaemia (Blood and lymphatic system disorders) | 1 | 10 | 1
Lymphopenia (Blood and lymphatic system disorders) | 6 | 8 | 8
Hypothyroidism (Endocrine disorders) | 24 | 10 | 0
Vision Blurred (Eye disorders) | 5 | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 91 | 87 | 11
Nausea (Gastrointestinal disorders) | 26 | 36 | 22
Constipation (Gastrointestinal disorders) | 26 | 26 | 16
Vomiting (Gastrointestinal disorders) | 10 | 25 | 7
Stomatitis (Gastrointestinal disorders) | 14 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 7 | 11 | 2
Oral Pain (Gastrointestinal disorders) | 8 | 5 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 7 | 4
Dry Mouth (Gastrointestinal disorders) | 5 | 7 | 1
Faecal Incontinence (Gastrointestinal disorders) | 7 | 0 | 0
Fatigue (General disorders) | 65 | 72 | 30
Oedema Peripheral (General disorders) | 17 | 16 | 8
Asthenia (General disorders) | 5 | 12 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 9 | 3
Urinary Tract Infection (Infections and infestations) | 5 | 8 | 2
Contusion (Injury, poisoning and procedural complications) | 7 | 10 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 6 | 5
Platelet Count Decreased (Investigations) | 3 | 21 | 9
White Blood Cell Count Decreased (Investigations) | 0 | 15 | 7
Weight Decreased (Investigations) | 6 | 14 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 13 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 13 | 2
Aspartate Aminotransferase Increased (Investigations) | 2 | 9 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 28 | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 12 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 10 | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 10 | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 7 | 3
Headache (Nervous system disorders) | 35 | 40 | 24
Convulsion (Nervous system disorders) | 17 | 9 | 7
Dizziness (Nervous system disorders) | 13 | 7 | 4
Aphasia (Nervous system disorders) | 12 | 4 | 3
Lethargy (Nervous system disorders) | 5 | 7 | 3
Hemiparesis (Nervous system disorders) | 4 | 4 | 5
Confusional State (Psychiatric disorders) | 10 | 6 | 1
Depression (Psychiatric disorders) | 7 | 10 | 3
Anxiety (Psychiatric disorders) | 5 | 9 | 3
Insomnia (Psychiatric disorders) | 9 | 9 | 8
Agitation (Psychiatric disorders) | 8 | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 10 | 4 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 39 | 36 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 16 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 1
Rash (Skin and subcutaneous tissue disorders) | 13 | 10 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 9 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 9 | 1 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 6 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 4
Hypertension (Vascular disorders) | 64 | 57 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.